CLINICAL TRIAL: NCT06324136
Title: Validation, Implementation, and Cost-analysis of a Strategy for Personalized Diagnosis of Rare Kidney Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Paola Romagnani, Professor, MD, PhD, Meyer Children's Hospital IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KIDNEY-PNRR
Record Dates: First submitted 2024-03-01; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rare kidney diseases (Experimental): Patients with rare kidney diseases
  Interventions: Diagnostic Test: Implementation of the diagnostic algorithm

INTERVENTIONS:
Diagnostic Test: Implementation of the diagnostic algorithm — Patients will be selected based on specific clinical criteria and referred to the tertiary center for genetic testing. All selected patients will undergo genetic testing by whole-exome sequencing (WES), followed by in silico analysis for an extended panel of genes associated with kidney diseases. The results of genetic testing will be evaluated by a multidisciplinary team of experts to establish conclusive diagnosis.

SUMMARY:
Chronic kidney disease (CKD) affects about 10% of the world population, with high morbidity and mortality. Genetic kidney diseases are increasingly recognized across all age groups and represent over 20% of all the causes of CKD. Accurate diagnosis allows necessary and unnecessary diagnostic procedures to be defined, avoids unnecessary treatments, improves prognosis prediction, identifies other family members for genetic counseling, and defines risks for living donor kidney transplantation. The research group coordinated by the Principal Investigator has recently developed an algorithm for the genetic diagnosis in pediatric and adult patients with CKD. The application of this personalized diagnostic algorithm on a local study led to a global diagnostic yield of 70%, suggesting that this strategy has the potential to substantially improve the diagnostic approach to patients with rare kidney disorders. The aim of this study is to validate and implement these results by extending its application in a multicentric study involving nephrology units that are referral centers for rare kidney diseases at national level.

ELIGIBILITY:
Inclusion Criteria:

* proteinuria and/or hematuria in the absence of immune deposits on renal biopsy or immune-mediated glomerulopathy resistant to treatment (e.g., steroids, immunosuppressive drugs);
* family history of kidney diseases and/or consanguinity;
* extrarenal involvement;
* ultrasound evidence of at least two cysts in each kidney or hyperechogenic kidneys or nephrocalcinosis;
* persistent metabolic abnormalities (metabolic acidosis or alkalosis without kidney function impairment; calcium phosphate metabolism abnormalities) after exclusion of secondary causes;
* availability of clinical information.
* signed informed consent form

Exclusion Criteria:

* Refusal by the patient, parents, or legal guardian to provide informed consent.

Ages: 0 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Implementation of a diagnostic algorithm for personalized diagnosis of rare kidney diseases | From enrollment of the first patient until the end of the study (up to 24 months)
  The previously established diagnostic algorithm for rare kidney diseases will be extended to out-of-region centers with a multicenter study design.
  This outcome will be assessed as diagnostic rate of the algorithm, i.e., number of conclusive genetic diagnosis/number of patients enrolled.

SECONDARY OUTCOMES:
Analysis of the functional role of variant of unknown clinical significance (VUS) | Form enrollment until the last follow up visit (up to 12 months)
  Analysis of the functional role of VUS identified by WES by in vitro functional studies and 3D-organ-on-a-chip models obtained by patients-specific urine-derived renal progenitor cells (u-RPC) cultures
Identification of immunological and/or structural factors in genetic and nongenetic forms. | Form enrollment until the last follow up visit (up to 12 months)
  Identification of immunological and/or structural factors in genetic and nongenetic forms.
  In particular, the investigators will assess:
  - the presence of anti-nephrin antibodies on serum samples and/or kidney biopsy of patients (performed for diagnostic purposes)
Cost-effectiveness of the diagnostic algorithm. | From enrollment of the last patient until the end of the study (up to 24 months)
  A modeled cost-effectiveness analysis (including direct and indirect medical costs) will be performed to compare the proposed diagnostic algorithm with the current standard-of-care.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Meyer Children's Hospital IRCCS, Florence
  - Azienda Ospedaliero Universitaria Vanvitelli, Napoli
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo

IPD SHARING:
Plan to Share IPD: No